CLINICAL TRIAL: NCT00934076
Title: Phase I Study of Erlotinib (Tarceva) in Combination With AT-101 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Tarceva and AT-101 for Patients With Advanced Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was never activated
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Ascenta Therapeutics (Industry)
Responsible Party: Francisco Robert, M.D., University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F090218006; UAB 0831 (Other: Institutional study protocol number)
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2011-01

CONDITIONS: Carcinoma, Non Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; gossypol acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AT-101 plus Erlotinib (Experimental): Subjects will begin study treatment at 150 mg of erlotinib taken once daily in a continuous regimen expressed in 3 week cycles.
  Subjects will begin treatment with oral AT-101 at 40 mg twice daily for 3 days of each 3 week cycle on an outpatient basis.
  Interventions: Drug: Tarceva plus AT-101

INTERVENTIONS:
Drug: Tarceva plus AT-101 — 150 mg of Tarceva taken once daily in a continuous regimen expressed in 3 week cycles.
  Oral AT-101 at 40 mg twice daily for 3 days of each 3 week cycle on an outpatient basis.

SUMMARY:
The purpose of this study the safety and effectiveness of oral AT-101 when given with the standard dose of erlotinib (Tarceva)to patients who are older that 18 and who have advanced non-small cell lung cancer, who have relapsed or progressed on prior platinum-based chemotherapy.

It is proposed that the effects of AT-101 may improve the clinical benefit of erlotinib in patients with advanced NSCLC.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of death in the United States as well as worldwide. It is estimated that approximately 215,020 new cases of lung cancer will be diagnosed in the United States in 2008, with approximately 161,840 deaths (1). The great majority of the lung cancers are grouped as non small cell lung cancer (NSCLC), and only 13% as small cell lung cancer. Most patients with NSCLC present with advanced disease (55% with stage IIIB or IV). The overall median survival of patients with advanced NSCLC treated with first line platinum based doublets is less than 12 months (8 10 months) with a 1 year and 2 year survival of 33% and 11%, respectively (2-4). Agents targeting epidermal growth factor receptor (EGFR), matrix metalloproteinase, farnesyl transferase, protein kinase C and retinoic X receptor have so far shown no survival benefit in combination with chemotherapy in advanced NSCLC (5-10).

More recently, 2 trials have shown clinical evidence of anti tumor activity with the addition of bevacizumab to first line chemotherapy in patients with advanced NSCLC (11,12). The pivotal study (EGOC 4599) responsible for the approval of bevacizumab in combination with carboplatin plus paclitaxel in selective patients with advanced non squamous cell lung cancers demonstrated a 2 month improvement in the median survival (12.3 months versus 10.3 months), and a higher objective response rate (12).

Patients with disease progression on or after first line therapy may be candidates for second line chemotherapy with either docetaxel or pemetrexed, which results in a modest improvement in survival. More recently, 2 EGFR tyrosine kinase inhibitors (TKIs), gefitinib and erlotinib, have been approved for second and third line therapy in advanced NSCLC (13,14). The effect on overall survival in genotypically uncharacterized patients was observed with erlotinib (BR21 trial), but not with gefitinib (ISEL trial), contributing to the withdrawal of gefitinib from the United States, and the approval of erlotinib as second and third line therapy in NSCLC irrespective of tumor genotype (15).

It is proposed that the effects of AT-101 on the downstream signaling pathways of the EGFR, particularly inhibition of the anti-apoptotic members Bcl-2 family of proteins, may provide an opportunity to improve the clinical benefit of erlotinib in patients with advanced NSCLC.

The safety of the combination of erlotinib with AT-101 has not been assessed. It is therefore proposed that a phase I study be performed using standard (FDA approved) dose of erlotinib (150 mg/day) with an effective dose of AT-101 (40 mg twice daily for 3 days) of a 3 week cycle.

ELIGIBILITY:
Inclusion Criteria:

* Pathological proven diagnosis of NSCLC with positive EGFR status by immunohistochemistry. Patients will be considered as positive if greater than 10% of the tumor cells are positively stained by the EGFR pharmDX assay kit.
* Disease that is locally advanced, metastatic, or recurrent.
* Prior treatment with 1 or 2 chemotherapy regimens, including a platinum based regimen for advanced disease (stage IIIB with malignant pleural effusion or stage IV).
* Evidence of unidimensionally measurable disease as per Response Evaluation Criteria in Solid Tumors [RECIST].
* Radiographic evidence of disease progression during or following previous chemotherapy treatment.
* Formalin fixed, paraffin embedded tumor tissue from the initial diagnoses will be obtained.
* Male or female, 19 years of age or older.
* ECOG performance status 0 2.
* Resolution of all acute toxic effects of prior therapy or surgical procedures (except for alopecia).
* Bisphosphonate therapy for bone metastases is allowed; however, treatment must be initiated prior to the first dose of therapy. Prophylactic use of bisphosphonates in patients without bone disease, except for the treatment of osteoporosis, is not permitted.
* Ability to swallow and retain oral medication.
* Adequate organ function as defined by the following criteria:

  * Hemoglobin >9.0 g/dL.
  * Absolute neutrophil count (ANC) >1500/μL.
  * Platelet >100,000/μL.
  * Serum creatinine <1.75 × ULN.
  * Serum albumin >3.0 g/dL.
  * Total serum bilirubin <1.5 × ULN.
  * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) <2.5 × ULN, or AST and ALT <5 × ULN if liver function abnormalities are due to underlying malignancy
* Signed and dated informed consent indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Males and non-pregnant, non-lactating females age 19 years or older.

Exclusion Criteria:

* Prior treatment with >2 systemic chemotherapy based regimens for advanced disease (stages IIIB/IV).
* Prior treatment with any EGFR inhibitors (TK inhibitor or monoclonal antibody).
* Symptomatic brain metastases or spinal cord compression; subjects will be eligible after adequate treatment (radiotherapy, surgery) and having stable disease not requiring steroids.
* Diagnosis of any second malignancy within the last 3 years, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma that has been adequately treated.
* Any significant acute or chronic medical (e.g., gastrointestinal complications, myocardial infarction, unstable angina, congestive heart failure, cerebrovascular accident, infection, metabolic complications, etc.) or psychiatric conditions that would impart, in the judgment of the investigator, excess risk associated with study participation, or study drug administration.
* Known human immunodeficiency virus (HIV) infection.
* Current treatment on other therapeutic clinical trials.
* Known hypersensitivity to gossypol, its enantiomers, or its excipients.
* Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.
* Patients with symptomatic hypercalcemia or hypercalcemia that is > grade 2.
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel are excluded. Subjects with ulcerative colitis, inflammatory bowel disease, or partial or complete small bowel obstruction are also excluded.
* Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test within 3 days prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability of erlotinib plus AT-101 | Assessment of toxicity will be performed on day 15 of the first cycle, and then on day 1 of every cycle of treatment.

SECONDARY OUTCOMES:
Evaluation of efficacy for erlotinib plus AT-101 using the binary outcome "alive without progression at 6 months (AWOP6)" as a secondary endpoint. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, M.D., Principal Investigator — University of Alabama at Birmingham